CLINICAL TRIAL: NCT00300066
Title: Prediction Equations for Glomerular Filtration Rate in Children Based on Serum Cystatin C and Body Cell Mass
Brief Title: Assessment of Serum Cystatin C as a Marker of Kidney Function in Children
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Trine Borup Andersen, MD, Department of Nuclear Medicine
Other Study IDs: VN-20050065MCH
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Kidney Disease
Keywords: Glomerular Filtration Rate; Serum Cystatin C; Body Composition; bioelectrical impedance spectroscopy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to assess serum cystatin C as a marker of kidney function (glomerular filtration rate, GFR) in children aged 2-14. The individual production rate and possible extra renal elimination of cystatin C based on body composition data is included to develop new algorithms to estimate GFR.

Furthermore, day-to-day variation on serum cystatin C is investigated.

DETAILED DESCRIPTION:
Today, children's kidney function (glomerular filtration rate, GFR) can be monitored by two methods:

1. indirectly by serum creatinine, or
2. directly by injection of a radioactive substance followed by several blood samples.

The first method is inaccurate with many drawbacks, whereas the latter is precise but time-consuming and unpleasant for the child. Therefore, there is a need for a new method for investigating GFR in children.

Serum cystatin C is a small protein that is produced with a constant rate in all nucleated cells in the body. It meets many of the characteristics of an ideal marker of GFR because of the way it is excreted in the kidneys. However, earlier studies have not proven serum cystatin C to be convincingly better than serum creatinine. Why? If there is considerable extra renal elimination, serum cystatin C alone isn't enough to estimate GFR. Therefore, the individual production rate and possible extra renal elimination of cystatin C are included in this study. To assess these factors, the children are submitted to bioelectrical impedance spectroscopy (BIS) to estimate their body composition, including body cell mass as cystatin C is produced in all nucleated cells. To validate the BIS data, dual energy x-ray absorptiometry (DEXA) will be conducted on 100 of the included children.

Based on serum cystatin C and the individual, age-corrected extra renal elimination rate of cystatin C, new algorithms to calculate GFR can be developed.

Furthermore, day-to-day variation in serum cystatin C and BIS data, which is expected to be low, is investigated in 100 of the included children.

Hypotheses:

1. Day-to-day variation on serum cystatin C is low.
2. Serum cystatin C raises parallel to falling GFR with time, which means that serum cystatin C can be used to monitor changes in kidney function in each patient.
3. Based on body composition, regression analysis and serum cystatin C values, GFR can be estimated in children aged 2-14.
4. GFR calculated as stated above is a more precise measurement of kidney function and changes in kidney function than GFR estimated from serum creatinine.
5. Data of body composition estimated by BIS do not deviate from data estimated by DEXA
6. Day-to-day variation in data for body composition measured by BIS is low.

The project includes 200 children aged 2-14 who are referred for routine examination of GFR in two Departments of Nuclear Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-14 years referred for GFR measurement by 51-CrEDTA

Exclusion Criteria:

* GFR measurement by capillary technique
* Immune compromising treatment
* Previous kidney transplant
* Hypo- or hyperthyroidism
* Increased C-reactive protein (CRP)
* Rheumatoid arthritis
* Ascites
* Pacemaker (only exclusion for BIS and DEXA)

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 2-14 years referrede for GFR measurement
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trine B Andersen, MD, Principal Investigator — University Hospital of Aarhus
Locations (2):
- Denmark (2):
  - Department of Nuclear Medicine, University Hospital Aarhus, Skejby, Aarhus, Brendstrupgaardsvej 100
  - Department of Clinical Physiology, University Hospital of Aarhus, Aalborg, Aalborg, Hobrovej 18-22